CLINICAL TRIAL: NCT06930118
Title: An Exploratory Study Investigating the Combination of Chidamide, Regorafenib, Plus Iparomlimab and Tuvonralimab for the Treatment of Drug-esistant and Efractory Dvanced Colorectal Cancer
Brief Title: The Aim of This Study is to Assess the Efficacy and Safety of Chidamide, Regorafenib in Combination With Iparomlimab and Tuvonralimab for the Treatment of Advanced Colorectal Cancer in Third-line Therapy and Subsequent Lines.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Apical-vict
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Advanced Colorectal Cancer in the Third-line Treatment and Beyond; pMMR/MSS Advanced Colorectal Cancer
Keywords: advanced colorectal cancer
MeSH Terms: interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; regorafenib

STUDY DESIGN:
Intervention Model Description: The aim of this study is to assess the efficacy and safety of the combination regimen of chidamide, regorafenib, and iparomlimab/tuvonralimab in patients with advanced colorectal cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- the combination regimen of chidamide, regorafenib, and iparomlimab/tuvonralimab (Experimental)
  Interventions: Drug: chidamide, regorafenib, and iparomlimab/tuvonralimab

INTERVENTIONS:
Drug: chidamide, regorafenib, and iparomlimab/tuvonralimab — All patients were treated with the following regimen: Chidamide: 30mg per dose, twice a week; Regorafenib: 80mg per dose, once a day, orally for 3 weeks, followed by a 1-week rest, and repeated every 4 weeks; Iparomlimab/Tuvonralimab: 5mg/kg, once every 3 weeks, intravenous infusion.

SUMMARY:
Patients with advanced colorectal cancer, particularly those of the pMMR/MSS type, exhibit suboptimal therapeutic responses in the third-line and subsequent treatments. The efficacy of the existing standard treatment regimens is highly restricted. In the CORRECT study, the median overall survival (OS) of regorafenib was 6.4 months, the median progression-free survival (PFS) was 1.9 months, and the objective response rate (ORR) was 1%. In the CONCUR study targeting the Asian population, the median OS of the regorafenib group was 8.8 months, the median PFS was 3.2 months, and the ORR was 4%. In the FRESCO study, the median OS of fruquintinib was 9.3 months, the median PFS was 3.7 months, and the ORR was 4.7%. In the TERRA study, the median OS of trifluridine/tipiracil (TAS-102) was 7.8 months, the median PFS was 2.0 months, and the ORR was 1.1%. The SUNLIGHT study explored the combined treatment modality of TAS-102 plus bevacizumab, where the median OS of the combined regimen was 10.8 months, the median PFS was 5.6 months, and the ORR was 6.1%. Evidently, the therapeutic efficacy of advanced colorectal cancer in the third-line and beyond has plateaued. In recent years, fundamental research has discovered that epigenetic regulation significantly synergizes with anti-angiogenesis and immune checkpoint inhibition therapy. Small-scale clinical explorations have also indicated favorable efficacy and clinical prospects, warranting further investigation. Hence, we contemplate employing the combination of chidamide, regorafenib, and iparomlimab/tuvonralimab to investigate its efficacy and safety in the treatment of advanced colorectal cancer in the third-line and beyond, and to explore novel breakthroughs for refractory colorectal cancer after multiple lines of treatment.

The aim of this study is to assess the efficacy and safety of the combination regimen of chidamide, regorafenib, and iparomlimab/tuvonralimab in patients with advanced colorectal cancer in the third-line and beyond. The study will be conducted at Shanghai Changzheng Hospital. The study drugs, including chidamide, regorafenib, and iparomlimab/tuvonralimab, are all commercially available in China.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced colorectal adenocarcinoma confirmed by histology or cytology;
* Those who have experienced disease progression or are intolerant to treatment after receiving ≥ 2 lines of systemic standard therapy;
* Patients must have at least one measurable lesion (according to RECIST 1.1 criteria);
* Patients who have received local radiotherapy at least 3 weeks before the first drug treatment are eligible for inclusion; however, the lesions evaluated by RECIST must not be within the radiotherapy field;
* Patients must be at least 18 years old;
* Performance status ECOG score of 0-1;
* Expected survival ≥ 12 weeks;
* Patients must have the ability to understand and voluntarily sign the written informed consent form;
* Women of childbearing age must have a negative pregnancy test within 7 days before the start of treatment. During the study period, both the patient and the patient's spouse must take contraceptive measures.

Exclusion Criteria:

* Patients who have undergone major surgery or suffered severe trauma within 4 weeks prior to the first dose of the study drug;
* Patients with hypersensitivity to any component of the study protocol;
* Patients planning to conceive or who are pregnant;
* Patients with brain metastases and an inability to accurately describe their condition;
* Patients who have experienced any of the following diseases within 6 months prior to the start of the study treatment: myocardial infarction, severe/unstable angina pectoris, NYHA class 2 or higher congestive heart failure, uncontrolled arrhythmia, etc.;
* Abnormal laboratory tests:

Absolute neutrophil count (ANC) < 1,500/mm3; Platelet count < 75,000/mm3; Total bilirubin > 1.5 times the upper limit of normal; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 2.5 times the upper limit of normal (for patients with liver metastases > 5 times the upper limit of normal); Creatinine > 1.5 times the upper limit of normal;

* Patients who have had other cancers (except advanced colorectal cancer) within 5 years prior to the start of this study treatment. Cervical carcinoma in situ, cured basal cell carcinoma and bladder epithelial tumors are excluded;
* Patients with a history of drug abuse, drug addiction, or alcohol dependence;
* Patients without legal capacity or with limited civil capacity;
* Other conditions that the investigator deems inappropriate for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate, ORR | From enrollment to the end of treatment at 8 weeks
  CR+PR

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Second Affiliated Hospital of Naval Medical University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751
- [Result] Ellis L, Hammers H, Pili R. Targeting tumor angiogenesis with histone deacetylase inhibitors. Cancer Lett. 2009 Aug 8;280(2):145-53. doi: 10.1016/j.canlet.2008.11.012. Epub 2008 Dec 25. PMID 19111391
- [Result] Thurn KT, Thomas S, Moore A, Munster PN. Rational therapeutic combinations with histone deacetylase inhibitors for the treatment of cancer. Future Oncol. 2011 Feb;7(2):263-83. doi: 10.2217/fon.11.2. PMID 21345145
- [Result] Grothey A, Van Cutsem E, Sobrero A, Siena S, Falcone A, Ychou M, Humblet Y, Bouche O, Mineur L, Barone C, Adenis A, Tabernero J, Yoshino T, Lenz HJ, Goldberg RM, Sargent DJ, Cihon F, Cupit L, Wagner A, Laurent D; CORRECT Study Group. Regorafenib monotherapy for previously treated metastatic colorectal cancer (CORRECT): an international, multicentre, randomised, placebo-controlled, phase 3 trial. Lancet. 2013 Jan 26;381(9863):303-12. doi: 10.1016/S0140-6736(12)61900-X. Epub 2012 Nov 22. PMID 23177514
- [Result] Heinemann V, von Weikersthal LF, Decker T, Kiani A, Vehling-Kaiser U, Al-Batran SE, Heintges T, Lerchenmuller C, Kahl C, Seipelt G, Kullmann F, Stauch M, Scheithauer W, Hielscher J, Scholz M, Muller S, Link H, Niederle N, Rost A, Hoffkes HG, Moehler M, Lindig RU, Modest DP, Rossius L, Kirchner T, Jung A, Stintzing S. FOLFIRI plus cetuximab versus FOLFIRI plus bevacizumab as first-line treatment for patients with metastatic colorectal cancer (FIRE-3): a randomised, open-label, phase 3 trial. Lancet Oncol. 2014 Sep;15(10):1065-75. doi: 10.1016/S1470-2045(14)70330-4. Epub 2014 Jul 31. PMID 25088940
- [Result] Suenaga M, Mizunuma N, Matsusaka S, Shinozaki E, Ozaka M, Ogura M, Chin K, Yamaguchi T. A phase I/II study of biweekly capecitabine and irinotecan plus bevacizumab as second-line chemotherapy in patients with metastatic colorectal cancer. Drug Des Devel Ther. 2015 Mar 16;9:1653-62. doi: 10.2147/DDDT.S80449. eCollection 2015. PMID 25834402
- [Result] Masi G, Salvatore L, Boni L, Loupakis F, Cremolini C, Fornaro L, Schirripa M, Cupini S, Barbara C, Safina V, Granetto C, Fea E, Antonuzzo L, Boni C, Allegrini G, Chiara S, Amoroso D, Bonetti A, Falcone A; BEBYP Study Investigators. Continuation or reintroduction of bevacizumab beyond progression to first-line therapy in metastatic colorectal cancer: final results of the randomized BEBYP trial. Ann Oncol. 2015 Apr;26(4):724-730. doi: 10.1093/annonc/mdv012. Epub 2015 Jan 18. PMID 25600568
- [Result] Cremolini C, Loupakis F, Antoniotti C, Lupi C, Sensi E, Lonardi S, Mezi S, Tomasello G, Ronzoni M, Zaniboni A, Tonini G, Carlomagno C, Allegrini G, Chiara S, D'Amico M, Granetto C, Cazzaniga M, Boni L, Fontanini G, Falcone A. FOLFOXIRI plus bevacizumab versus FOLFIRI plus bevacizumab as first-line treatment of patients with metastatic colorectal cancer: updated overall survival and molecular subgroup analyses of the open-label, phase 3 TRIBE study. Lancet Oncol. 2015 Oct;16(13):1306-15. doi: 10.1016/S1470-2045(15)00122-9. Epub 2015 Aug 31. PMID 26338525
- [Result] Li J, Qin S, Xu R, Yau TC, Ma B, Pan H, Xu J, Bai Y, Chi Y, Wang L, Yeh KH, Bi F, Cheng Y, Le AT, Lin JK, Liu T, Ma D, Kappeler C, Kalmus J, Kim TW; CONCUR Investigators. Regorafenib plus best supportive care versus placebo plus best supportive care in Asian patients with previously treated metastatic colorectal cancer (CONCUR): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2015 Jun;16(6):619-29. doi: 10.1016/S1470-2045(15)70156-7. Epub 2015 May 13. PMID 25981818
- [Result] Giannakis M, Mu XJ, Shukla SA, Qian ZR, Cohen O, Nishihara R, Bahl S, Cao Y, Amin-Mansour A, Yamauchi M, Sukawa Y, Stewart C, Rosenberg M, Mima K, Inamura K, Nosho K, Nowak JA, Lawrence MS, Giovannucci EL, Chan AT, Ng K, Meyerhardt JA, Van Allen EM, Getz G, Gabriel SB, Lander ES, Wu CJ, Fuchs CS, Ogino S, Garraway LA. Genomic Correlates of Immune-Cell Infiltrates in Colorectal Carcinoma. Cell Rep. 2016 Apr 26;15(4):857-865. doi: 10.1016/j.celrep.2016.03.075. Epub 2016 Apr 14. PMID 27149842
- [Result] Jones PA, Issa JP, Baylin S. Targeting the cancer epigenome for therapy. Nat Rev Genet. 2016 Sep 15;17(10):630-41. doi: 10.1038/nrg.2016.93. PMID 27629931
- [Result] Orillion A, Hashimoto A, Damayanti N, Shen L, Adelaiye-Ogala R, Arisa S, Chintala S, Ordentlich P, Kao C, Elzey B, Gabrilovich D, Pili R. Entinostat Neutralizes Myeloid-Derived Suppressor Cells and Enhances the Antitumor Effect of PD-1 Inhibition in Murine Models of Lung and Renal Cell Carcinoma. Clin Cancer Res. 2017 Sep 1;23(17):5187-5201. doi: 10.1158/1078-0432.CCR-17-0741. Epub 2017 Jul 11. PMID 28698201
- [Result] Turajlic S, Litchfield K, Xu H, Rosenthal R, McGranahan N, Reading JL, Wong YNS, Rowan A, Kanu N, Al Bakir M, Chambers T, Salgado R, Savas P, Loi S, Birkbak NJ, Sansregret L, Gore M, Larkin J, Quezada SA, Swanton C. Insertion-and-deletion-derived tumour-specific neoantigens and the immunogenic phenotype: a pan-cancer analysis. Lancet Oncol. 2017 Aug;18(8):1009-1021. doi: 10.1016/S1470-2045(17)30516-8. Epub 2017 Jul 7. PMID 28694034
- [Result] O'Neil BH, Wallmark JM, Lorente D, Elez E, Raimbourg J, Gomez-Roca C, Ejadi S, Piha-Paul SA, Stein MN, Abdul Razak AR, Dotti K, Santoro A, Cohen RB, Gould M, Saraf S, Stein K, Han SW. Safety and antitumor activity of the anti-PD-1 antibody pembrolizumab in patients with advanced colorectal carcinoma. PLoS One. 2017 Dec 28;12(12):e0189848. doi: 10.1371/journal.pone.0189848. eCollection 2017. PMID 29284010
- [Result] Li J, Qin S, Xu RH, Shen L, Xu J, Bai Y, Yang L, Deng Y, Chen ZD, Zhong H, Pan H, Guo W, Shu Y, Yuan Y, Zhou J, Xu N, Liu T, Ma D, Wu C, Cheng Y, Chen D, Li W, Sun S, Yu Z, Cao P, Chen H, Wang J, Wang S, Wang H, Fan S, Hua Y, Su W. Effect of Fruquintinib vs Placebo on Overall Survival in Patients With Previously Treated Metastatic Colorectal Cancer: The FRESCO Randomized Clinical Trial. JAMA. 2018 Jun 26;319(24):2486-2496. doi: 10.1001/jama.2018.7855. PMID 29946728
- [Result] Xu RH, Muro K, Morita S, Iwasa S, Han SW, Wang W, Kotaka M, Nakamura M, Ahn JB, Deng YH, Kato T, Cho SH, Ba Y, Matsuoka H, Lee KW, Zhang T, Yamada Y, Sakamoto J, Park YS, Kim TW. Modified XELIRI (capecitabine plus irinotecan) versus FOLFIRI (leucovorin, fluorouracil, and irinotecan), both either with or without bevacizumab, as second-line therapy for metastatic colorectal cancer (AXEPT): a multicentre, open-label, randomised, non-inferiority, phase 3 trial. Lancet Oncol. 2018 May;19(5):660-671. doi: 10.1016/S1470-2045(18)30140-2. Epub 2018 Mar 16. PMID 29555258
- [Result] Xu J, Kim TW, Shen L, Sriuranpong V, Pan H, Xu R, Guo W, Han SW, Liu T, Park YS, Shi C, Bai Y, Bi F, Ahn JB, Qin S, Li Q, Wu C, Ma D, Lin D, Li J. Results of a Randomized, Double-Blind, Placebo-Controlled, Phase III Trial of Trifluridine/Tipiracil (TAS-102) Monotherapy in Asian Patients With Previously Treated Metastatic Colorectal Cancer: The TERRA Study. J Clin Oncol. 2018 Feb 1;36(4):350-358. doi: 10.1200/JCO.2017.74.3245. Epub 2017 Dec 7. PMID 29215955
- [Result] Aderka D, Stintzing S, Heinemann V. Explaining the unexplainable: discrepancies in results from the CALGB/SWOG 80405 and FIRE-3 studies. Lancet Oncol. 2019 May;20(5):e274-e283. doi: 10.1016/S1470-2045(19)30172-X. PMID 31044725
- [Result] Bekaii-Saab TS, Ou FS, Ahn DH, Boland PM, Ciombor KK, Heying EN, Dockter TJ, Jacobs NL, Pasche BC, Cleary JM, Meyers JP, Desnoyers RJ, McCune JS, Pedersen K, Barzi A, Chiorean EG, Sloan J, Lacouture ME, Lenz HJ, Grothey A. Regorafenib dose-optimisation in patients with refractory metastatic colorectal cancer (ReDOS): a randomised, multicentre, open-label, phase 2 study. Lancet Oncol. 2019 Aug;20(8):1070-1082. doi: 10.1016/S1470-2045(19)30272-4. Epub 2019 Jun 28. PMID 31262657
- [Result] Chen EX, Jonker DJ, Loree JM, Kennecke HF, Berry SR, Couture F, Ahmad CE, Goffin JR, Kavan P, Harb M, Colwell B, Samimi S, Samson B, Abbas T, Aucoin N, Aubin F, Koski SL, Wei AC, Magoski NM, Tu D, O'Callaghan CJ. Effect of Combined Immune Checkpoint Inhibition vs Best Supportive Care Alone in Patients With Advanced Colorectal Cancer: The Canadian Cancer Trials Group CO.26 Study. JAMA Oncol. 2020 Jun 1;6(6):831-838. doi: 10.1001/jamaoncol.2020.0910. PMID 32379280
- [Result] Fukuoka S, Hara H, Takahashi N, Kojima T, Kawazoe A, Asayama M, Yoshii T, Kotani D, Tamura H, Mikamoto Y, Hirano N, Wakabayashi M, Nomura S, Sato A, Kuwata T, Togashi Y, Nishikawa H, Shitara K. Regorafenib Plus Nivolumab in Patients With Advanced Gastric or Colorectal Cancer: An Open-Label, Dose-Escalation, and Dose-Expansion Phase Ib Trial (REGONIVO, EPOC1603). J Clin Oncol. 2020 Jun 20;38(18):2053-2061. doi: 10.1200/JCO.19.03296. Epub 2020 Apr 28. PMID 32343640
- [Result] Que Y, Zhang XL, Liu ZX, Zhao JJ, Pan QZ, Wen XZ, Xiao W, Xu BS, Hong DC, Guo TH, Shen LJ, Fan WJ, Chen HY, Weng DS, Xu HR, Zhou PH, Zhang YZ, Niu XH, Zhang X. Frequent amplification of HDAC genes and efficacy of HDAC inhibitor chidamide and PD-1 blockade combination in soft tissue sarcoma. J Immunother Cancer. 2021 Feb;9(2):e001696. doi: 10.1136/jitc-2020-001696. PMID 33637599
- [Result] Wang F, He MM, Yao YC, Zhao X, Wang ZQ, Jin Y, Luo HY, Li JB, Wang FH, Qiu MZ, Lv ZD, Wang DS, Li YH, Zhang DS, Xu RH. Regorafenib plus toripalimab in patients with metastatic colorectal cancer: a phase Ib/II clinical trial and gut microbiome analysis. Cell Rep Med. 2021 Aug 27;2(9):100383. doi: 10.1016/j.xcrm.2021.100383. eCollection 2021 Sep 21. PMID 34622226
- [Result] Cousin S, Cantarel C, Guegan JP, Gomez-Roca C, Metges JP, Adenis A, Pernot S, Bellera C, Kind M, Auzanneau C, Le Loarer F, Soubeyran I, Bessede A, Italiano A. Regorafenib-Avelumab Combination in Patients with Microsatellite Stable Colorectal Cancer (REGOMUNE): A Single-arm, Open-label, Phase II Trial. Clin Cancer Res. 2021 Apr 15;27(8):2139-2147. doi: 10.1158/1078-0432.CCR-20-3416. Epub 2021 Jan 25. PMID 33495314
- [Result] Zhong M, Lin F, Jiang Y, Pan G, Tan J, Zhou H, Lai Q, Chen Q, Deng M, Zha J, Xu B. Therapeutic Interaction of Apatinib and Chidamide in T-Cell Acute Lymphoblastic Leukemia through Interference with Mitochondria Associated Biogenesis and Intrinsic Apoptosis. J Pers Med. 2021 Sep 29;11(10):977. doi: 10.3390/jpm11100977. PMID 34683119
- [Result] Garralda E, Sukari A, Lakhani NJ, Patnaik A, Lou Y, Im SA, Golan T, Geva R, Wermke M, de Miguel M, Palcza J, Jha S, Chaney M, Abraham AK, Healy J, Falchook GS. A first-in-human study of the anti-LAG-3 antibody favezelimab plus pembrolizumab in previously treated, advanced microsatellite stable colorectal cancer. ESMO Open. 2022 Dec;7(6):100639. doi: 10.1016/j.esmoop.2022.100639. Epub 2022 Dec 6. PMID 36493599
- [Result] Mettu NB, Ou FS, Zemla TJ, Halfdanarson TR, Lenz HJ, Breakstone RA, Boland PM, Crysler OV, Wu C, Nixon AB, Bolch E, Niedzwiecki D, Elsing A, Hurwitz HI, Fakih MG, Bekaii-Saab T. Assessment of Capecitabine and Bevacizumab With or Without Atezolizumab for the Treatment of Refractory Metastatic Colorectal Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2022 Feb 1;5(2):e2149040. doi: 10.1001/jamanetworkopen.2021.49040. PMID 35179586
- [Result] Tabernero J, Grothey A, Arnold D, de Gramont A, Ducreux M, O'Dwyer P, Tahiri A, Gilberg F, Irahara N, Schmoll HJ, Van Cutsem E. MODUL cohort 2: an adaptable, randomized, signal-seeking trial of fluoropyrimidine plus bevacizumab with or without atezolizumab maintenance therapy for BRAFwt metastatic colorectal cancer. ESMO Open. 2022 Oct;7(5):100559. doi: 10.1016/j.esmoop.2022.100559. Epub 2022 Aug 24. PMID 36029653
- [Result] Andre T, Lonardi S, Wong KYM, Lenz HJ, Gelsomino F, Aglietta M, Morse MA, Van Cutsem E, McDermott R, Hill A, Sawyer MB, Hendlisz A, Neyns B, Abdullaev S, Memaj A, Lei M, Dixon M, Kopetz S, Overman MJ. Nivolumab plus low-dose ipilimumab in previously treated patients with microsatellite instability-high/mismatch repair-deficient metastatic colorectal cancer: 4-year follow-up from CheckMate 142. Ann Oncol. 2022 Oct;33(10):1052-1060. doi: 10.1016/j.annonc.2022.06.008. Epub 2022 Jun 25. PMID 35764271
- [Result] Guo Y, Zhang W, Ying J, Zhang Y, Pan Y, Qiu W, Fan Q, Xu Q, Ma Y, Wang G, Guo J, Su W, Fan S, Tan P, Wang Y, Luo Y, Zhou H, Li J. Phase 1b/2 trial of fruquintinib plus sintilimab in treating advanced solid tumours: The dose-escalation and metastatic colorectal cancer cohort in the dose-expansion phases. Eur J Cancer. 2023 Mar;181:26-37. doi: 10.1016/j.ejca.2022.12.004. Epub 2022 Dec 13. PMID 36628898
- [Result] Fakih M, Raghav KPS, Chang DZ, Larson T, Cohn AL, Huyck TK, Cosgrove D, Fiorillo JA, Tam R, D'Adamo D, Sharma N, Brennan BJ, Wang YA, Coppieters S, Zebger-Gong H, Weispfenning A, Seidel H, Ploeger BA, Mueller U, Oliveira CSV, Paulson AS. Regorafenib plus nivolumab in patients with mismatch repair-proficient/microsatellite stable metastatic colorectal cancer: a single-arm, open-label, multicentre phase 2 study. EClinicalMedicine. 2023 Apr 6;58:101917. doi: 10.1016/j.eclinm.2023.101917. eCollection 2023 Apr. PMID 37090438
- [Result] Fakih M, Sandhu J, Lim D, Li X, Li S, Wang C. Regorafenib, Ipilimumab, and Nivolumab for Patients With Microsatellite Stable Colorectal Cancer and Disease Progression With Prior Chemotherapy: A Phase 1 Nonrandomized Clinical Trial. JAMA Oncol. 2023 May 1;9(5):627-634. doi: 10.1001/jamaoncol.2022.7845. PMID 36892833
- [Result] Prager GW, Taieb J, Fakih M, Ciardiello F, Van Cutsem E, Elez E, Cruz FM, Wyrwicz L, Stroyakovskiy D, Papai Z, Poureau PG, Liposits G, Cremolini C, Bondarenko I, Modest DP, Benhadji KA, Amellal N, Leger C, Vidot L, Tabernero J; SUNLIGHT Investigators. Trifluridine-Tipiracil and Bevacizumab in Refractory Metastatic Colorectal Cancer. N Engl J Med. 2023 May 4;388(18):1657-1667. doi: 10.1056/NEJMoa2214963. PMID 37133585
- [Result] Han B, Zheng R, Zeng H, Wang S, Sun K, Chen R, Li L, Wei W, He J. Cancer incidence and mortality in China, 2022. J Natl Cancer Cent. 2024 Feb 2;4(1):47-53. doi: 10.1016/j.jncc.2024.01.006. eCollection 2024 Mar. PMID 39036382
- [Result] Wang F, Jin Y, Wang M, Luo HY, Fang WJ, Wang YN, Chen YX, Huang RJ, Guan WL, Li JB, Li YH, Wang FH, Hu XH, Zhang YQ, Qiu MZ, Liu LL, Wang ZX, Ren C, Wang DS, Zhang DS, Wang ZQ, Liao WT, Tian L, Zhao Q, Xu RH. Combined anti-PD-1, HDAC inhibitor and anti-VEGF for MSS/pMMR colorectal cancer: a randomized phase 2 trial. Nat Med. 2024 Apr;30(4):1035-1043. doi: 10.1038/s41591-024-02813-1. Epub 2024 Mar 4. PMID 38438735